CLINICAL TRIAL: NCT05856162
Title: Early Intervention to Promote Cardiovascular Health of Mothers and Children at Northwestern University
Brief Title: Early Intervention to Promote Cardiovascular Health of Mothers and Children
Acronym: ENRICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Darius Tandon, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00216961
Record Dates: First submitted 2023-04-04; First posted 2023-05-12 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Intervention (Experimental): Participants randomized to this arm will receive the full ENRICH pilot which will consist of content on diet, physical activity, sleep, stress/mental health, and tobacco cessation. They will also receive usual home visiting services.
  Interventions: Behavioral: ENRICH pilot intervention (full intervention)
- Diet/Physical Activity Intervention (Active Comparator): Participants randomized to this arm will receive the partial ENRICH pilot which will consist of content on diet and physical activity. They will also receive usual home visiting services.
  Interventions: Behavioral: ENRICH pilot intervention (partial intervention: only diet and physical activity)
- Control (No Intervention): Participants randomized to this arm will receive no ENRICH intervention content. They will only receive usual home visiting services.

INTERVENTIONS:
Behavioral: ENRICH pilot intervention (full intervention) — The full ENRICH pilot intervention will consist of content related to diet, physical activity, stress/mental health, sleep, tobacco cessation, and child health. The investigators will use an adapted version of the Mothers and Babies stress management intervention to address mental health, an adapted version of the HEALTH curriculum to address diet/physical activity, and an adapted version of the INSIGHT curriculum to address child health.
  Arms: Full Intervention
Behavioral: ENRICH pilot intervention (partial intervention: only diet and physical activity) — The partial ENRICH intervention will focus only on diet and physical activity.
  Arms: Diet/Physical Activity Intervention

SUMMARY:
The goal of this clinical trial is to examine whether a multi-component intervention delivered during pregnancy and after delivery can improve the cardiovascular health of pregnant individuals enrolled in home visiting programs, as well as their offspring's cardiovascular health. The main questions it aims to answer are:

1. Does a multi-component intervention improve cardiovascular health of pregnant individuals and new mothers enrolled in home visiting programs?
2. Does a multi-component intervention improve cardiovascular health of the offspring of pregnant individuals/new mothers enrolled in home visiting programs?

Participants receiving the multi-component intervention will receive content on promoting cardiovascular health delivered by their home visitor and asynchronously. All participants will be asked to complete assessments at baseline, 2-month follow-up, and 4-month follow-up. The investigators will compare whether pregnant individuals and new mothers randomized to the intervention group, and their offspring, exhibit better cardiovascular health than pregnant individuals and new mothers randomized to the control group.

DETAILED DESCRIPTION:
Poor cardiovascular health (CVH) is highly prevalent among pregnant individuals and is associated with adverse maternal and offspring outcomes. As CVH is already suboptimal by early adolescence, early-life interventions are needed. Interventions conducted in the community by trusted programs have the potential to improve CVH risk factors among perinatal individuals and their children. Home Visiting (HV) programs are trusted maternal and child health providers in diverse US communities, especially among low-income families.

This project is part of the National Heart Lung and Blood Institute (NHLBI) Early Intervention to Promote Cardiovascular Health of Mothers and Children (ENRICH) consortium. Northwestern University is one seven clinical centers part of the ENRICH consortium. This project is funded via a UG3/UH3 mechanism in which during the UG3 period each clinical center is responsible for conducting a pilot study to inform the development of a common protocol that will be used across all seven clinical centers during the UH3 phase. This clinicaltrials.gov entry describes the pilot RCT protocol.

The pilot study will use a randomized controlled trial (RCT) longitudinal design. Forty individuals randomized to the intervention arm will receive usual home visiting services along with the ENRICH intervention. Ten individuals randomized to the control arm will receive usual home visiting without the ENRICH intervention. Among the individuals randomized to the intervention condition, 20 (50%) will receive the entire ENRICH intervention while the other 20 will receive only diet and physical activity content. The varying levels of intervention dosage is being delivered to assess acceptability and feasibility of a more- and less-intensive version of the intervention. Components of the intervention are described below. Assessments will be conducted at baseline, 2-month follow-up, and 4-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years old
* Pregnant or with child < 3 months of age
* Enrolled in a Healthy Families America or Parents as Teachers home visiting program in Illinois or or Indiana

Exclusion Criteria:

* Individuals pregnant with twins (or higher order gestation)
* Individuals who have a fetus with a known chromosomal abnormality

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in diet assessed via the Mediterranean Eating Pattern for Americans Questionnaire | Change in eating patterns between baseline, 2 month follow-up, and 4 month follow-up
  Use of Mediterranean/DASH diet. The MEPA range is from 0-16 with higher scores indicating greater use of a Mediterranean diet
Change in maternal physical activity assessed via the International Physical Activity Questionnaire (IPAQ) | Change in physical activity between baseline, 2 month follow-up, and 4 month follow-up
  Engagement in physical activity. The IPAQ contains 12 questions with responses scored to create low, moderate, and high physical activity categories

SECONDARY OUTCOMES:
Change in maternal depression symptoms assessed via the Edinburgh Postnatal Depression Scale (EPDS) | Change in maternal depression between baseline, 2 month follow-up, and 4 month follow-up
  Depressive symptoms. The EPDS is a 10-item scale with a range of 0-30. Higher scores reflect more depressive symptomatology

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States